CLINICAL TRIAL: NCT07164872
Title: Neoadjuvant Chemotherapy Combined With Preoperative Radiotherapy for Locally Advanced Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, JIN JING, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS2025-6-1
Record Dates: First submitted 2025-08-07; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; preoperative radiotherapy; pCR
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preoperative radiotherapy (Experimental): whole breast irradiation of the affected side ± chest wall + regional lymph node drainage area irradiation: whole breast ± chest wall + supraclavicular and internal mammary regional lymph node drainage area 40.05Gy/152.67Gy/ day per session, axillary regional lymph node drainage area 37.5Gy/15f,2.5Gy/ per session
  Interventions: Radiation: preoperative radiotherapy

INTERVENTIONS:
Radiation: preoperative radiotherapy — preoperative radiotherapy

SUMMARY:
Approximately 20% of breast cancer patients in our country are in the locally advanced stage. The relatively low overall survival rate, high recurrence rate and distant metastasis risk of these patients significantly affect the therapeutic efficacy and survival. Preoperative radiotherapy is a treatment option for many tumors. It is recommended to administer radiotherapy and systemic chemotherapy before surgery to enhance preoperative tumor downstaging, eliminate micrometastatic lesions and improve overall survival rate. Preoperative radiotherapy combined with chemotherapy for breast cancer patients further shrinks the tumor, increases the probability of breast preservation, and may also eliminate the need for axillary lymph node dissection, thereby improving the quality of life of patients. Pathological complete response (pCR) not only helps with subsequent surgery but also has significant advantages in improving survival rate. Neoadjuvant radiotherapy is also one of the treatment options for reducing tumor stage, but it has not been widely applied to breast cancer patients. Among breast cancer subtypes, Luminal type accounts for 50-70%, among which HR+ HER2- breast cancer patients have poor efficacy from neoadjuvant chemotherapy and pCR rate is below 5-10%. Triple-negative breast cancer accounts for 15-20% of all breast cancer subtypes. It has the characteristics of poor differentiation, strong invasiveness, earlier and more frequent recurrence and metastasis. The efficacy of traditional neoadjuvant chemotherapy has approached its limit. This study aims to explore the efficacy and safety of neoadjuvant radiotherapy for locally advanced breast cancer.

DETAILED DESCRIPTION:
Approximately one fifth of the patients in China have non-metastatic locally advanced breast cancer. Due to their relatively low overall survival rate, high recurrence rate, and risk of distant metastasis, this significantly affects the therapeutic efficacy and survival of the patients. Preoperative neoadjuvant radiotherapy is a common treatment option for many tumors (such as esophageal cancer, rectal cancer, soft tissue sarcoma, etc.), by advancing radiotherapy and systemic chemotherapy to before surgery to enhance preoperative treatment for tumor downstaging and early elimination of micrometastatic lesions to improve overall survival rate. In breast cancer patients, preoperative radiotherapy combined with chemotherapy has the opportunity to further shrink the tumor, increase the probability of breast preservation, and possibly avoid axillary lymph node dissection, thereby improving the quality of life of the patients. Pathological complete response (pCR) not only helps subsequent surgical treatment but also has significant advantages in improving survival rate, significantly improving the overall prognosis of patients. Neoadjuvant radiotherapy is also one of the treatment options for reducing the stage. However, this combination has not been widely applied to breast cancer patients yet and further clinical research is needed. Among all breast cancers, Luminal-type breast cancer accounts for 50-70%, among which patients with HR+HER2- type breast cancer have poor efficacy of neoadjuvant chemotherapy and the pCR rate is usually below 5-10%. Triple-negative breast cancer accounts for 15-20% of all breast cancer subtypes, characterized by poor differentiation, strong invasiveness, earlier and more frequent recurrence and metastasis. The efficacy of traditional neoadjuvant chemotherapy has approached its limit and the pCR rate hovers around 35%. This study aims to explore the pCR rate, effectiveness and safety of preoperative chemotherapy combined with preoperative medium-dose fractionated radiotherapy in patients with locally advanced HR+HER2- type and triple-negative breast cancer, to improve the overall survival of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. The pathological diagnosis was invasive breast cancer.
2. cT3-4, cN1-2, M0 (according to the 8th edition of the AJCC Cancer Staging Manual), molecular typing is Luminal type (HER2-) or triple-negative type. The volume of the primary lesion did not decrease by more than 50% after 2 cycles of neoadjuvant chemotherapy.
3. Generally in good condition (KPS score > 70), organ functions are tolerable, and there are no severe complications due to poor control.
4. Acceptable for magnetic resonance imaging scan
5. Have the conditions for follow-up
6. Sign the informed consent form

Exclusion Criteria:

1. gestation period
2. Simultaneous bilateral breast cancer
3. History of chest wall radiotherapy
4. Active connective tissue disease
5. Inflammatory breast cancer
6. Excessive breast volume (>600ml), BMI > 30
7. diabetes
8. Positive lymph nodes in the upper and lower regions of the clavicle and the internal mammary region
9. Using immunotherapy drugs such as PD-1/PD-L1

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete respons | 8-12 weeks
  pathological complete

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-11-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT07164872/Prot_000.pdf